CLINICAL TRIAL: NCT00885053
Title: The Effect of Acute and Short-term Intervention With Fish Oil on Overweight Subjects - Focus on Inflammation
Brief Title: Fish Oil and Inflammation in Overweight Subjects
Acronym: ADIPOMEGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Trine Madsen / MD, Department of Cardiology, Aalborg Hospital, Aarhus University Hospital, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ADIPOMEGA
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2009-12

CONDITIONS: Overweight
Keywords: Inflammation; Fatty acids, Omega 3; Leukotrienes; Adiponectin; Adipose tissue; RNA, Messenger
MeSH Terms: conditions — Overweight; Inflammation | interventions — Fish Oils; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish oil (Experimental)
  Interventions: Dietary Supplement: fish oil
- Olive oil (Placebo Comparator)
  Interventions: Dietary Supplement: olive oil

INTERVENTIONS:
Dietary Supplement: fish oil — Capsules. Approximately 1000 mg n-3 PUFA daily. One day + 6 weeks
  Arms: Fish oil
Dietary Supplement: olive oil — Capsules. Approximately 1 g olive oil daily. One day + 6 weeks
  Arms: Olive oil

SUMMARY:
The aim of this study is to investigate the effects of acute and short-term intervention with fish oil on inflammatory markers in overweight subjects.

DETAILED DESCRIPTION:
Being overweight is associated with metabolic syndrome, cardiovascular disease, and diabetes mellitus (type 2). Adipose tissue can be regarded as an active organ, which produces an array of inflammatory mediators. This creates a state of chronic low-grade inflammation. Inflammation has been proven to be a key element in the development of atherosclerotic plaques.

The marine n-3 polyunsaturated fatty acids (PUFAs) have beneficial effects on cardiovascular disease. These effects are partly attributed to the anti-inflammatory effect of the n-3 PUFAs.

Previous studies have shown an anti-inflammatory effect of n-3 PUFAs in overweight subjects, but the studies have been conducted with a high daily dose of n-3 PUFA. We want to examine the effect of a lower dose of 1 g n-3 PUFA/day (the dose recommended by the Danish Heart Foundation).

The study is randomized, placebo-controlled and double blinded. Fifty subjects aged 30 - 75 years (postmenopausal women; waist circumference > 80 cm and men; waist circumference > 94 cm) will be included.

Blood samples and fatty tissue biopsies will be collected at baseline, after 1 day and after 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference ≥ 80 cm (females) or ≥ 94 cm (males)
* Postmenopausal (females)

Exclusion Criteria:

* Daily intake of fish oil capsules
* Daily intake of NSAIDs
* HbA1c ≥ 8%
* Serum creatinine ≤ 30 mL/min
* Chronic inflammatory disease
* Other serious illness
* Inability to informed consent

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To assess the effect of 1 g/day of n-3 polyunsaturated fatty acids on inflammatory markers | After 1 day and after 6 weeks intervention

SECONDARY OUTCOMES:
To assess effect of 1 g n-3 polyunsaturated fatty acids (daily dose) on the fatty acid profile of plasma, leucocytes and adipose tissue. | After 1 day and 6 after weeks of intervention
To assess the effect of 1g n-3 polyunsaturated fatty acids (daily dose) on the gene expression profile (mRNA) - especially genes involved in encoding the inflammatory response. | After 1 day and 6 after weeks of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg Hospital, Aarhus University Hospital, Aalborg, Denmark

REFERENCES:
- [Background] Hajer GR, van Haeften TW, Visseren FL. Adipose tissue dysfunction in obesity, diabetes, and vascular diseases. Eur Heart J. 2008 Dec;29(24):2959-71. doi: 10.1093/eurheartj/ehn387. Epub 2008 Sep 5. PMID 18775919
- [Background] Balkau B, Deanfield JE, Despres JP, Bassand JP, Fox KA, Smith SC Jr, Barter P, Tan CE, Van Gaal L, Wittchen HU, Massien C, Haffner SM. International Day for the Evaluation of Abdominal Obesity (IDEA): a study of waist circumference, cardiovascular disease, and diabetes mellitus in 168,000 primary care patients in 63 countries. Circulation. 2007 Oct 23;116(17):1942-51. doi: 10.1161/CIRCULATIONAHA.106.676379. PMID 17965405
- [Background] Libby P, Ridker PM, Maseri A. Inflammation and atherosclerosis. Circulation. 2002 Mar 5;105(9):1135-43. doi: 10.1161/hc0902.104353. PMID 11877368
- [Background] Calder PC. n-3 polyunsaturated fatty acids, inflammation, and inflammatory diseases. Am J Clin Nutr. 2006 Jun;83(6 Suppl):1505S-1519S. doi: 10.1093/ajcn/83.6.1505S. PMID 16841861
- [Background] Schmidt EB, Arnesen H, de Caterina R, Rasmussen LH, Kristensen SD. Marine n-3 polyunsaturated fatty acids and coronary heart disease. Part I. Background, epidemiology, animal data, effects on risk factors and safety. Thromb Res. 2005;115(3):163-70. doi: 10.1016/j.thromres.2004.09.006. PMID 15617737
- [Background] Schmidt EB, Arnesen H, Christensen JH, Rasmussen LH, Kristensen SD, De Caterina R. Marine n-3 polyunsaturated fatty acids and coronary heart disease: Part II. clinical trials and recommendations. Thromb Res. 2005;115(4):257-62. doi: 10.1016/j.thromres.2004.09.007. No abstract available. PMID 15668184
- [Background] Browning LM, Krebs JD, Moore CS, Mishra GD, O'Connell MA, Jebb SA. The impact of long chain n-3 polyunsaturated fatty acid supplementation on inflammation, insulin sensitivity and CVD risk in a group of overweight women with an inflammatory phenotype. Diabetes Obes Metab. 2007 Jan;9(1):70-80. doi: 10.1111/j.1463-1326.2006.00576.x. PMID 17199721
- [Background] Kris-Etherton PM, Harris WS, Appel LJ; AHA Nutrition Committee. American Heart Association. Omega-3 fatty acids and cardiovascular disease: new recommendations from the American Heart Association. Arterioscler Thromb Vasc Biol. 2003 Feb 1;23(2):151-2. doi: 10.1161/01.atv.0000057393.97337.ae. No abstract available. PMID 12588750